CLINICAL TRIAL: NCT01100281
Title: Neuropsychological and Anatomical Study of Concept Formation in Frontal Patients
Brief Title: Prefrontal Cortex and Abstract Thinking
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C09-29
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Abstract Thinking; Concept Formation
Keywords: prefrontal cortex
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PSP (Progressive supranuclear palsy)
  Interventions: Behavioral: Neuropsychological examination; Other: MRI
- FTD (Frontotemporal lobar degenerative)
  Interventions: Behavioral: Neuropsychological examination; Other: MRI
- Alzheimer's disease
  Interventions: Behavioral: Neuropsychological examination; Other: MRI

INTERVENTIONS:
Behavioral: Neuropsychological examination — Examination including especially concept formation
Other: MRI — MRI performed in T1-weighted three dimensional sequence

SUMMARY:
The capacity of concept formation is not well understood, even if a link is supposed with the functioning of the frontal lobes.

Our aim is to better understand the cognitive mechanisms underlying this function and to try to correlate the performance with atrophy of the frontal lobe in neurodegenerative diseases involving this region (frontotemporal lobar degeneration and progressive supranuclear palsy).

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* MMSE> 20
* No contra indication to MRI

Exclusion Criteria:

* MMSE<20

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups including : PSP, FTD, AD
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2010-04; Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Inserm U 975, Paris, France